CLINICAL TRIAL: NCT03004885
Title: Enhanced Lung Protective Ventilation for ARDS Patients With PrismaLung
Acronym: PROVAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient CO2 removal obtained with the PrismaLung membrane oxygenator
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, MD, MSc, Hôpital Européen Marseille
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A01523-48
Record Dates: First submitted 2016-12-14; First posted 2016-12-29 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Minimal Distension (Experimental): Tidal volume 4 ml/kg PBW and PEEP based on the ARDSNet PEEP/FiO2 table (ARMA) + ECCO2R
  Interventions: Device: PrismaLung
- Maximal Recruitment (Experimental): Tidal volume 4 ml/kg PBW and PEEP adjusted to maintain plateau pressure between 23 - 25 cmH2O + ECCO2R
  Interventions: Device: PrismaLung
- Standard (Active Comparator): Tidal volume 6 ml/kg PBW and PEEP based on the ARDSNet PEEP/FiO2 table (ARMA) without ECCO2R
  Interventions: Device: PrismaLung

INTERVENTIONS:
Device: PrismaLung — Low flow Extracorporeal CO2 removal using a 0.32 m² membrane oxygenator

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) still remains associated with a mortality rate of 30 - 45 % despite improvement in mechanical ventilation. Driving pressure, defined as the difference between the end-inspiratory and the end-expiratory airway pressure, appears as an important factor contributing to mortality in patients with the ARDS. In patients already receiving a conventional tidal volume of 6 ml/kg predicted body weight (PBW), a driving pressure ≥ 14 cmH2O increases the risk of death in the hospital. One mean to lower the driving pressure is to decrease the tidal volume such that from 6 to 4 ml/kg predicted body weight. However, this strategy promotes hypercarbia by reducing the alveolar ventilation, providing the respiratory rate is constant. In this setting, implementing an extracorporeal CO2 removal (ECCO2R) therapy may offset the associated hypercarbia. The investigators have previously demonstrated that combining a membrane oxygenator within an hemofiltration circuit provides efficacious low flow ECCO2R on a renal replacement therapy monitor. In this study, we thought to investigate the efficacy of the PrismaLung stand-alone therapy. Using a PrismaFlex monitor and a HP-X circuit, a neonatal membrane oxygenator (PrismaLung) is used to provide decarboxylation without renal replacement therapy. The study will consist in three periods:

* The first period will address the efficacy of the PrismaLung device at tidal volume of 6 and 4 ml/kg PBW using an off-on-off design.
* The second part of the study will investigate the effect of varying the sweep gas flow and the mixture of the sweep gas on the CO2 removal rate (random order).
* The third part will compare three ventilatory strategies applied in a cross-over design :

  1. Minimal distension: Tidal volume 4 ml/kg PBW and positive end-expiratory pressure (PEEP) based on the ARDSNet PEEP/FiO2 table (ARMA).
  2. Maximal recruitment: 4 ml/kg PBW and PEEP adjusted to maintain a plateau pressure between 23 - 25 cmH2O.
  3. Standard: Tidal volume 6 ml/kg and PEEP based on the ARDSNet PEEP/FiO2 table (ARMA).

Each strategies will be apply in a random order for a duration of 22 hours. Pulmonary inflammatory and fibrosis pathway will be assess before and after each period using bronchoalveolar lavage (BAL) samples. Systemic inflammatory cytokines will also be investigate. Main measurements will include respiratory mechanics, transpulmonary pressure, work of breathing, end-expiratory lung volume and tidal ventilation using electrical impedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* ARDS moderate or severe (Berlin criteria)
* Onset < 48 h
* Driving pressure ≥ 14 cmH2O

Exclusion Criteria:

* Lack of consent or social protection
* Chronic respiratory failure (requiring Oxygen or NIPPV)
* Severe hypoxemia: PaO2/FIO2 < 100 with PEEP ≥ 18 cmH2O AND FIO2 = 1
* Acute Renal Failure requiring RRT
* DNR order or death expected within the next 72 hours
* Planned surgery or out-of-ICU transportation expected within the next 72 hours
* Heparin allergy
* Contraindication to jugular vein catheterization
* Intracranial Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change in PaCO2 | 15 min after initiation of ECCO2R (PrismaLung) at tidal volume of 4 ml/kg PBW (during the first part of the study).
  20 % decrease in PaCO2 after initiation of ECCO2R (PrismaLung) at tidal volume of 4 ml/kg PBW versus 4 ml/kg PBW without ECCO2R.

SECONDARY OUTCOMES:
PaCO2 | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Arterial blood gas
CO2 removal rate | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Using both the blood side and the gas side equation
Respiratory mechanics work of breathing | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Using oesophageal ballon (NutriVent catheter) and FluxMed monitor (MBMed)
Transpulmonary pressure | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Using oesophageal ballon (NutriVent catheter) and FluxMed monitor (MBMed)
Work of breathing | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Using oesophageal ballon (NutriVent catheter) and FluxMed monitor (MBMed)
EIT | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Electrical Impedance Tomography using BB² (Swisstom)
EELV | q15 min during part 1 and part 2 of the study. In the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  End expiratory Lung volume using nitrogen wash-in wash-out method (Engstrom GE)
Plasma Cytokines | Only in the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Elisa using plasma samples
Pulmonary Cytokines | Only in the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  Elisa using BAL samples
Pulmonary Type III Procollagen | Only in the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  RIA using plasma and BAL samples
Pulmonary Inflammatory and Fibrotic pathway | Only in the third part, measurement at baseline, 1 hour and 22 hours in each arm.
  mRNA

OTHER OUTCOMES:
Plasma Free Hemoglobin | q24 h, up to 72 h
Haptoglobin | q24 h, up to 72 h
Lacticodéshydrogenase (LDH) | q24 h, up to 72 h
schizocytes | q24 h, up to 72 h
Bilirubin | q24 h, up to 72 h

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Europeen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Allardet-Servent J, Castanier M, Signouret T, Soundaravelou R, Lepidi A, Seghboyan JM. Safety and Efficacy of Combined Extracorporeal CO2 Removal and Renal Replacement Therapy in Patients With Acute Respiratory Distress Syndrome and Acute Kidney Injury: The Pulmonary and Renal Support in Acute Respiratory Distress Syndrome Study. Crit Care Med. 2015 Dec;43(12):2570-81. doi: 10.1097/CCM.0000000000001296. PMID 26488219